CLINICAL TRIAL: NCT05699044
Title: Prevalence, Characteristics and Prognosis of Transthyretin Amyloidosis in Patients With New-onset Advanced AV-block - A National Screening Study
Brief Title: Screening of ATTRwt in Patient With Advanced AV-Block Undergoing Pacemaker Implantation
Acronym: ATTRAB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Steen Hvitfeldt Poulsen (Other)
Responsible Party: Sponsor-Investigator, Steen Hvitfeldt Poulsen, Prof. Poulsen, Aarhus University Hospital Skejby
Organization: Aarhus University Hospital Skejby (Other)
Other Study IDs: 1-10-72-53-22
Record Dates: First submitted 2022-10-04; First posted 2023-01-26 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Amyloid Cardiomyopathy; Block, AV
MeSH Terms: conditions — Amyloid Neuropathies, Familial; Atrioventricular Block

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Bloodtest
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Amyloidosis Screening: Patients fulfilling eligibility criteria will screened for Cardiac Amyloidosis.
  Interventions: Diagnostic Test: Amyloidosis screening (bloodtest, DPD-scintigraphy, potentially endomyocardial biopsy)

INTERVENTIONS:
Diagnostic Test: Amyloidosis screening (bloodtest, DPD-scintigraphy, potentially endomyocardial biopsy) — Bloodtest: Troponin I, NT-pro-BNP, electrolyte status, renal function, kampda/lambda free chain + ratio, M-komponent.
  DPD-scintigraphy. (Echocardiography)

SUMMARY:
The investigators will nationally investigate the prevalence of Transthyretin Amyloidosis wildtype (ATTRwt) in patients of ≥ 65 years with left ventricular hypertrophy who present with high degree atrioventricular block (AV-block) and are admitted for pacemaker implantation. The investigators aim to characterize the group of patients with positive screening of ATTR and compare the ATTRwt disease stage at time of diagnosis for patients identified with ATTR at screening with a control group of routinely clinically diagnosed ATTRwt patients.

ELIGIBILITY:
Inclusion Criteria:

* Men ≥65years or women ≥75years with unexplained AV-block with pacemaker indication, as decided per treating physician and presence of left ventricular hypertrophy ≥12mm.

Exclusion Criteria:

* Reversible causes for AV-block, som as AV-node disturbing medicament, ion-disturbances, hypothyroidism, hypoxia, ischemia, new heart surgery <1month, endocarditis.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients admitted for pacemakerimplantation with advanced AV-block fulfilling eligibility criteria as described.
Sampling Method: Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of ATTRwt in study cohort. | 3 years
  Number of participants with a diagnosis of ATTRwt in the study cohort based on DPD-scintigraphy or if necessary, a cardiac biopsy.

SECONDARY OUTCOMES:
Characteristics of patients with ATTRwt | 3 years
  Echocardiographic (Left ventricular (LV) wall thickness, LV cavity dimension, EF, GLS, diastolic function, Right Ventricular (RV) systolic function, valve disease) Biochemical profile (Troponin I, NT-pro-BNP, Renal Function (E-GFR) ), presence or history of spinal stenosis, carpal tunnel syndrome
Clinical Stage of time of diagnosis in patients with ATTRwt | 3 years
  Gilmore Staging
Number of heart-failure associated hospitalization among ATTRwt patients | 5 years
All-cause mortality among ATTRwt patients. | 5 year

CONTACTS AND LOCATIONS:
Overall Officials: Steen Poulsen, MD, Principal Investigator — Department of Cardiology, Aarhus University Hospital
Locations (1):
- Department of Cardiology, Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Undecided